CLINICAL TRIAL: NCT05513573
Title: A Randomized, Double-Blind, Multi-Center Phase II Clinical Study to Compare the Efficacy and Safety of HLX07 (Recombinant Anti-EGFR Humanized Monoclonal Antibody Injection) + Serplulimab (HLX10, Recombinant Anti-PD-1 Humanized Monoclonal Antibody) +Chemotherapy Versus Placebo + Serplulimab + Chemotherapy in First-Line Treatment of Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)
Brief Title: Phase II Clinical Study to Compare the Efficacy and Safety of HLX07 + Serplulimab +Chemotherapy Versus Placebo + Serplulimab + Chemotherapy in First-Line Treatment of Patients With Recurrent or Metastatic NPC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX07-NPC201
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Nasopharyngeal Carcinoma by AJCC V8 Stage
MeSH Terms: interventions — HLX07; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX07+HLX10+chemotherapy (Experimental)
  Interventions: Drug: HLX07; Drug: HLX10; Drug: chemotherapy
- Placebo+HLX10+chemotherapy (Experimental)
  Interventions: Drug: HLX10; Drug: placebo; Drug: chemotherapy

INTERVENTIONS:
Drug: HLX07 — 1500 mg, D1，Q3W
  Arms: HLX07+HLX10+chemotherapy
Drug: HLX10 — 300 mg, D1, up to 2 years,Q3W
Drug: placebo — 1500 mg, D1，Q3W
  Arms: Placebo+HLX10+chemotherapy
Drug: chemotherapy — gemcitabine 1000 mg/m2, D1,D8; cisplatin 80 mg/m2,D1；Q3W, up to 6 cycles

SUMMARY:
A Randomized, Double-Blind, Multi-Center Phase II Clinical Study to Compare the Efficacy and Safety of HLX07 (Recombinant Anti-EGFR Humanized Monoclonal Antibody Injection) + Serplulimab (HLX10, Recombinant Anti-PD-1 Humanized Monoclonal Antibody) +Chemotherapy Versus Placebo + Serplulimab + Chemotherapy in First-Line Treatment of Patients with Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical study; fully understand, be informed about the study, and have signed the informed consent form (ICF); be willing to follow and be able to complete all trial procedures.
2. Males or females aged ≥ 18 years at the time of signing the ICF.
3. Histologically or cytologically proven recurrent or metastastic NPC.
4. At least one measurable target lesion is assessed by the IRRC according to the RECIST v1.1 within 4 weeks prior to randomization.
5. An ECOG performance status score of 0-1 within 7 days prior to the first dose of the investigational product.
6. An expected survival period ≥ 12 weeks.

Exclusion Criteria:

1. Other active malignancies within 3 years prior to the first dose of investigational product. Localized tumors that have been cured such as superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, and breast cancer in situ are acceptable.
2. Patients who are going to receive or have received an organ or bone marrow transplant.
3. With uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage (monthly or more frequently).
4. With cerebrovascular accident, myocardial infarction, unstable angina, poorly controlled arrhythmia (including QTc intervals ≥ 450 ms for males and ≥ 470 ms for females) (QTc intervals are calculated by Fridericia formula) within half a year.
5. Class III to IV cardiac insufficiency according to New York Heart Association (NYHA) classification (Appendix 5) or an LVEF (left ventricular ejection fraction) < 50% by cardiac color Doppler.
6. Inadequately controlled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg).
7. With human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 weeks
  Objective response rate (ORR) (assessed by the IRRC according to the RECIST v1.1 criteria)

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 14 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC and INV according to the RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No